CLINICAL TRIAL: NCT01978171
Title: Prediction of Everolimus-induced Interstitial Lung Disease in Breast Cancer Patients; Maximizing Efficacy by Reducing Toxicity
Brief Title: Prediction of Everolimus-induced Interstitial Lung Disease
Acronym: PREVENT
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCNONCO201302
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2017-09

CONDITIONS: Breast Neoplasms
Keywords: breast neoplasms; everolimus; interstitial lung disease; pneumonitis
MeSH Terms: conditions — Breast Neoplasms; Lung Diseases, Interstitial; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, skin biopsies, broncho-alveolar lavage fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- breast cancer patients: Postmenopausal women with estrogen receptor (ER) positive advanced breast cancer whose disease is refractory to non steroidal aromatase inhibitors, and are eligible for treatment with exemestane and everolimus.

SUMMARY:
The investigators will determine which factors are predictive for the development and severity of everolimus-induced interstitial lung disease and will develop a prediction model based on these risk factors.

DETAILED DESCRIPTION:
In this study the investigators will prospectively investigate pulmonary adverse events during treatment with everolimus. The investigators will distinguish the following everolimus-induced pulmonary adverse events: pulmonary infection, everolimus-induced airway disease and everolimus-induced interstitial lung disease (ILD). The investigators will investigate the predictive value of pneumoproteins, everolimus exposure, pulmonary function tests, four distinct radiological patterns, baseline patient characteristics and the development of skin toxicity or oral mucositis for the development and severity of everolimus-induced ILD.

ELIGIBILITY:
Inclusion Criteria:

* Adult women with metastatic or locally advanced breast cancer not amenable to curative treatment by surgery or radiotherapy.
* Histological or cytological confirmation of estrogen-receptor positive (ER+) breast cancer
* Postmenopausal women
* Radiological or clinical evidence of recurrence or progression on last systemic therapy prior to enrollment
* Resistance to treatment with a non-steroidal aromatase inhibitor
* Serum platelets ≥ 100x10E9/l
* Everolimus dose adjustment is recommended for patients with hepatic impairment (Child-Pugh A/B/C)
* Performance status ECOG 0 - 2 (Karnofsky index: 60 - 100)

Exclusion Criteria:

* Patients with a HER2-overexpressing tumor
* Known hypersensitivity to mTOR inhibitors, e.g. sirolimus (rapamycin).
* Patients with a known history of HIV seropositivity or hepatitis B or C
* Uncontrolled diabetes mellitus
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with estrogen receptor (ER) positive advanced breast cancer whose disease is refractory to non steroidal aromatase inhibitors, and are eligible for treatment with exemestane and everolimus.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2014-05; Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
predictive factors of everolimus-induced ILD | six months
  Find the correlation between:
  * pneumoproteins
  * everolimus exposure
  * pulmonary function tests
  * four distinct radiological patterns of 1.0mm CT slices of the lungs
  * baseline patient characteristics
  * the development and grade of everolimus-induced skin toxicity and oral mucositis
  and the development and grade of everolimus-induced ILD

SECONDARY OUTCOMES:
temporal relation pneumoproteins and ILD | six months
  Analyze the temporal relationship between a decrease in pulmonary function or the occurrence of new radiological pulmonary abnormalities and an increase in the level of pneumoproteins
pathophysiology of everolimus-induced ILD | six months
  Investigate which immunological changes (cytokines, T-cells, dendritic cells) are observed in peripheral blood, skin biopsies and bronchoalveolar lavage fluid of patients with everolimus-induced toxicity
relation ILD and exposure and outcome | six months
  Define the correlation between everolimus-induced ILD on the one hand and everolimus exposure (as per AUC0-24h) on day 14) and outcome (time to progression, as determined by treating physician) on the other hand

CONTACTS AND LOCATIONS:
Overall Officials: Carla van Herpen, MD, PhD, Principal Investigator — Radboud university medical center, department of medical oncology; Nielka van Erp, PharmD, PhD, Principal Investigator — Radboud university medical center, department of Pharmacy
Locations (2):
- Netherlands (2):
  - Antonius Ziekenhuis, Nieuwegein
  - Radboud university medical center, Nijmegen

REFERENCES:
- [Derived] Willemsen AECAB, Tol J, van Erp NP, Jonker MA, de Boer M, Meek B, de Jong PC, van Moorsel C, Gerritsen WR, Grutters JC, van Herpen CML. Prospective Study of Drug-induced Interstitial Lung Disease in Advanced Breast Cancer Patients Receiving Everolimus Plus Exemestane. Target Oncol. 2019 Aug;14(4):441-451. doi: 10.1007/s11523-019-00656-2. PMID 31325105